CLINICAL TRIAL: NCT06258278
Title: Clinical Results of Arthroscopic-Assisted Lower Trapezius Tendon Transfer for Massive, Irreparable Rotator Cuff Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Research asistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iayas7
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Massive Irreparable Rotator Cuff Tears
Keywords: Irreparable Rotator Cuff Tears; Tendon Transfer; Massive Rotator Cuff Tears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Massive Irreparable Rotator Cuff Tears (Experimental): Patients scheduled for arthroscopically assisted lower trapezius transfer due to irreparable massive rotator cuff tears
  Interventions: Procedure: Arthroscopic-assisted lower trapezius tendon transfer surgery

INTERVENTIONS:
Procedure: Arthroscopic-assisted lower trapezius tendon transfer surgery — The procedure, conducted under general anesthesia, starts with diagnostic arthroscopy followed by excision of the posterior bursa and preparation of the rotator cuff footprint. Attention then shifts to harvesting the low trapezius tendon, accessed through a 10cm incision over the spina scapula. The tendon is detached, dissected, and released from adhesions, ensuring not to damage its pedicle. A fascia lata graft is harvested from the ipsilateral thigh and sutured to the low trapezius tendon in a continuous, locking manner to aid fixation on the humeral head. A subdeltoid tunnel is formed, and the graft is shuttled into the subacromial space and fixed at the bicipital groove and tuberculum majus with knotless anchors. The stability of fixation and mobility of the low trapezius muscle are verified, and the graft and tendon are sutured together with tension, with the arm held in 90° abduction and maximum external rotation.

SUMMARY:
This study aimed to describe a modified technique for arthroscopic-assisted transfer of the lower trapezius tendon in a selected group of patients with irreparable rotator cuff tears and to evaluate its short-term results.

DETAILED DESCRIPTION:
Patients scheduled for surgery will undergo evaluation one day before the surgical procedure and again at the six-month postoperative mark. Pain intensity will be assessed using the Visual Analog Scale (VAS), while shoulder function will be evaluated using both the University of California, Los Angeles (UCLA) Shoulder Score and the Constant-Murley Shoulder Score.

ELIGIBILITY:
Inclusion Criteria:

* patients with massive, chronic (>6 months), irreparable rotator cuff tears;
* patients with no concomitant irreparable subscapularis tears;
* patients who underwent a trial of at least 6-month period of conservative treatment with no benefit;
* patients with a stage 3 or greater degree of supraspinatus muscle fatty infiltration;

Exclusion Criteria:

* patients with glenohumeral arthritis;
* patients with adhesive capsulitis or passive joint motion restriction
* patients with neurologic deficits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | one day before surgery
  Pain intensity is assessed using the Visual Analog Scale (VAS). Patients are presented with a 10-centimeter horizontal line labeled with 'No Pain' at one end (scored as 0) and 'Worst Pain Imaginable' at the other end (scored as 10). Patients are instructed to mark on the line the point that represents their current level of pain. The distance from the 'No Pain' end to the patient's mark is measured to determine the pain score, with higher scores indicating greater pain intensity.
Pain intensity | 6 months after surgery
  Pain intensity is assessed using the Visual Analog Scale (VAS). Patients are presented with a 10-centimeter horizontal line labeled with 'No Pain' at one end (scored as 0) and 'Worst Pain Imaginable' at the other end (scored as 10). Patients are instructed to mark on the line the point that represents their current level of pain. The distance from the 'No Pain' end to the patient's mark is measured to determine the pain score, with higher scores indicating greater pain intensity.
Shoulder ability | one day before surgery
  The Constant-Murley score is used to evaluate shoulder function. This scoring system comprises four subscales: pain (scored out of 15 points), activities of daily living (scored out of 20 points), range of motion (scored out of 40 points), and strength (scored out of 25 points), totaling a maximum score of 100 points. Each subscale is assessed through a series of standardized maneuvers and patient-reported outcomes.
Shoulder ability | 6 months after surgery
  The Constant-Murley score is used to evaluate shoulder function. This scoring system comprises four subscales: pain (scored out of 15 points), activities of daily living (scored out of 20 points), range of motion (scored out of 40 points), and strength (scored out of 25 points), totaling a maximum score of 100 points. Each subscale is assessed through a series of standardized maneuvers and patient-reported outcomes.
Shoulder function | one day before surgery
  The University of California, Los Angeles (UCLA) Shoulder Rating Scale is utilized to evaluate shoulder function. This scoring system consists of a series of questions assessing pain level, function, active forward flexion, strength, and patient satisfaction. Each category is scored on a scale ranging from 0 to 10 or 0 to 5, with higher scores indicating better function and satisfaction
Shoulder function | 6 months after surgery
  The University of California, Los Angeles (UCLA) Shoulder Rating Scale is utilized to evaluate shoulder function. This scoring system consists of a series of questions assessing pain level, function, active forward flexion, strength, and patient satisfaction. Each category is scored on a scale ranging from 0 to 10 or 0 to 5, with higher scores indicating better function and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Ulunay Kanatlı, Principal Investigator — Gazi University; Furkan Aral, Study Chair — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No